CLINICAL TRIAL: NCT03463577
Title: An Observational, Retrospective Cohort Database Study to Assess the Safety of Boostrix (U.S. Formulation), a Reduced Tetanus, Diphtheria, Acellular Pertussis Vaccine (Tdap), Following Routine Immunization of Pregnant Women in the United States
Brief Title: The Safety of Boostrix Following Routine Immunization of Pregnant Women
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Kaiser Permanente (Other)
Responsible Party: Sponsor
Other Study IDs: 207221
Record Dates: First submitted 2018-03-06; First posted 2018-03-13 (Actual); Results first posted 2022-05-18 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Whooping Cough
Keywords: whooping cough, Boostrix, Tdap, safety, pregnancy, infants
MeSH Terms: conditions — Whooping Cough | interventions — Boostrix

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (6):
- Exposed cohort women-on or after 1st day of 27th week of pregnancy: This group consisted of pregnant women who received the Tdap vaccine (Boostrix) on or after the 1st day of the 27th week of pregnancy during the period January 1, 2018 to January 31, 2019 who were not vaccinated with any other Tdap vaccine at any other time during the pregnancy.
  Interventions: Other: Safety assessment following routine immunization with Boostrix
- Unexposed historical cohort women: This group consisted of women matched to Exposed cohort women-on or after 1st day of 27th week of pregnancy group and pregnant at least one day during the historical period between January 1, 2012-December 31, 2014 and did not receive any Tdap vaccine during the pregnancy.
  Interventions: Other: Safety assessment following routine immunization with Boostrix
- Exposed cohort women-before 1st day of 27th week of pregnancy: This group consisted of pregnant women who received the Tdap vaccine (Boostrix) before the 1st day of the 27th week of pregnancy during the period January 1, 2018-January 31, 2019 who were not vaccinated with any other Tdap vaccine at any other time during the pregnancy.
  Interventions: Other: Safety assessment following routine immunization with Boostrix
- Exposed cohort infants-on or after 1st day of 27th week of pregnancy: This group consisted of infants whose mothers belong to Exposed cohort women-on or after 1st day of 27th week of pregnancy group.
  Interventions: Other: Safety assessment following routine immunization with Boostrix
- Unexposed historical cohort infants: This group consisted of infants whose mothers belong to the Unexposed historical cohort women group.
  Interventions: Other: Safety assessment following routine immunization with Boostrix
- Exposed cohort infants-before 1st day of 27th week of pregnancy: This group consisted of infants whose mothers belong to the Exposed cohort women-before 1st day of 27th week of pregnancy group.
  Interventions: Other: Safety assessment following routine immunization with Boostrix

INTERVENTIONS:
Other: Safety assessment following routine immunization with Boostrix — Subject-level data was collected for pregnant women and their infants through the Electronic Health Records.

SUMMARY:
The purpose of this study was to assess the safety of Boostrix administered on or after the first day of the 27th week of pregnancy by conducting a post-marketing study that provided safety information to the public and healthcare providers. This was one of the largest cohorts of pregnant women vaccinated with Boostrix in the U.S. Through partnership between Kaiser Permanente Southern California (KPSC) and the sponsor, GlaxoSmithKline (GSK), information about the safety of maternal vaccination with Boostrix and maternal and infant adverse events (AEs) in a community setting was gained.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with prenatal care and continuous membership (allowing up to a 31-day gap) at KPSC between the 1st day of the 27th week of pregnancy and the index (vaccination) date.
* Exposed cohort (from the 27th week of gestation): Pregnant women vaccinated with Boostrix on or after the 1st day of the 27th week of pregnancy; who were not vaccinated with any other Tdap vaccine at any other time during the pregnancy in scope of this study.
* Unexposed cohort: Women matched to the exposed cohort and pregnant sometime during the approximate estimated period between January 1, 2012-December 31, 2014 and did not receive any Tdap vaccine during the pregnancy in scope of this study.

For the analysis of congenital anomalies among live births, at birth and through six months of age, the following additional inclusion criteria for infants will be applied:

* Live born
* Born in KPSC hospitals

Note: Pregnant women vaccinated with Boostrix during pregnancy before the 27th week of gestation, with membership at the date of vaccination, and who were not vaccinated with any other Tdap vaccine at any other time during the pregnancy in scope of this study will be part of a descriptive analysis (secondary objective).

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Pregnant women with prenatal care and continuous membership (allowing up to a 31-day gap) at KPSC between the 1st day of the 27th week of pregnancy and the index (vaccination) date.
Study Population: Pregnant women with prenatal care and continuous membership (allowing up to a 31-day gap) at KPSC between the 1st day of the 27th week of pregnancy and the index date
Sampling Method: Non-Probability Sample
Enrollment: 65783 (Actual)
Dates: Start 2018-04-13 (Actual); Primary Completion 2020-08-04 (Actual); Study Completion 2020-08-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Pasadena, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Florea A, Sy LS, Ackerson BK, Qian L, Luo Y, Becerra-Culqui T, Lee GS, Tian Y, Zheng C, Bathala R, Tartof SY, Campora L, Ceregido MA, Kuznetsova A, Poirrier JE, Rosillon D, Valdes L, Cheuvart B, Mesaros N, Meyer N, Guignard A, Tseng HF. Investigating Tetanus, Diphtheria, Acellular Pertussis Vaccination During Pregnancy and Risk of Congenital Anomalies. Infect Dis Ther. 2023 Feb;12(2):411-423. doi: 10.1007/s40121-022-00731-8. Epub 2022 Dec 15. PMID 36520325

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Data was collected for both pregnant women and their infants from Kaiser Permanente Southern California (KPSC) Electronic Health Records (EHR).
Pre-assignment Details: The study population for the first analysis includes pregnant women who received Tdap (Boostrix) vaccine on or after the first day of the 27th week of pregnancy (Exposed cohort-on or after 1st day of 27th week of pregnancy) and their infants, as well as the matched unexposed pregnant women and their infants (Unexposed historical cohort). A second analysis was performed on pregnant women who received the Tdap vaccine before the 1st day of the 27th week of pregnancy, and their infants.
Period: Overall Study
Arm/Group | Exposed Cohort women-on or After 1st Day of 27th Week of Pregnancy | Unexposed Historical Cohort Women | Exposed Cohort Women-before 1st Day of 27th Week of Pregnancy | Exposed Cohort infants-on or After 1st Day of 27th Week of Pregnancy | Unexposed Historical Cohort Infants | Exposed Cohort Infants-before 1st Day of 27th Week of Pregnancy
Started | 16606 | 16606 | 65 | 16350 | 16088 | 68
Completed | 16366 | 16166 | 65 | 16335 | 16071 | 68
Not Completed | 240 | 440 | 0 | 15 | 17 | 0
Not completed — Lost to Follow-up | 238 | 435 | 0 | 0 | 0 | 0
Not completed — With unknown pregnancy outcome | 0 | 5 | 0 | 0 | 0 | 0
Not completed — Maternal death | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Neonatal death | 0 | 0 | 0 | 15 | 17 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Exposed Cohort women-on or After 1st Day of 27th Week of Pregnancy | Unexposed Historical Cohort Women | Exposed Cohort Women-before 1st Day of 27th Week of Pregnancy | Exposed Cohort infants-on or After 1st Day of 27th Week of Pregnancy | Unexposed Historical Cohort Infants | Exposed Cohort Infants-before 1st Day of 27th Week of Pregnancy | Total
Number analyzed (Participants) | 16606 | 16606 | 65 | 16350 | 16088 | 68 | 65783
Age, Customized [Count of Participants; unit: Participants]
  0-1 year | 0 | 0 | 0 | 16350 | 16088 | 68 | 32506
  13 -51 year | 16606 | 16606 | 65 | 0 | 0 | 0 | 33277
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16606 | 16606 | 65 | 7950 | 7725 | 36 | 48988
  Male | 0 | 0 | 0 | 8400 | 8363 | 32 | 16795
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 2974 | 2974 | 14 | 0 | 0 | 0 | 5962
  Black | 1274 | 1274 | 5 | 0 | 0 | 0 | 2553
  Hispanic | 9689 | 9689 | 31 | 0 | 0 | 0 | 19409
  Asian | 2144 | 2144 | 10 | 0 | 0 | 0 | 4298
  Other-Unspecified | 525 | 525 | 5 | 16350 | 16088 | 68 | 33561

OUTCOME MEASURES:

1. Primary Outcome: Incidence Rate (Per 1000 Person-years) of Pre-specified Maternal Adverse Events for Exposed Cohort women-on or After 1st Day of 27th Week of Pregnancy and Unexposed Historical Cohort-women Groups
Description: The incidence rate (per 1000) of maternal adverse events was calculated as the total number of adverse events in the numerator and the total person-years at risk in the denominator. Every unexposed woman was assigned an index date that is determined by the number of days from pregnancy start to the Boostrix vaccination date of her matched exposed woman. The same number of days calculated in the exposed woman was added to the pregnancy start of the unexposed woman to identify her index date. The pre-specified maternal adverse events assessed were pre-eclampsia and eclampsia; Intra-uterine infections.
Time Frame: From date of Boostrix vaccination (Exposed cohort women-on or after 1st day of 27th week of pregnancy) or from an index date (Unexposed historical cohort women) until end of enrollment or pregnancy, whichever came first, up to 13 weeks
Population: The analysis was performed on all women from the Exposed cohort women-on or after 1st day of 27th week of pregnancy group and the Unexposed historical cohort women group, who met the eligibility criteria and for whom the event could be assessed.
Measure: Number (95% Confidence Interval); unit: Events per 1000 persons-year
Arm/Group | Exposed Cohort women-on or After 1st Day of 27th Week of Pregnancy | Unexposed Historical Cohort Women
Number analyzed (Participants) | 16606 | 16606
Events per 1000 persons-year
  Pre-eclampsia and eclampsia | 316.16 [296.24 to 337.42] | 219.00 [202.13 to 237.28]
  Intra-uterine infections | 292.53 [273.56 to 312.81] | 207.35 [191.12 to 224.95]
Statistical Analysis 1: Comparison: Exposed Cohort women-on or After 1st Day of 27th Week of Pregnancy vs Unexposed Historical Cohort Women; Demonstration of adjusted relative risk (RR) for pre-eclampsia and eclampsia in Exposed women cohort (on or after 1st day of 27th week of pregnancy) compared to Unexposed historical women cohort was less than 2 (non-inferiority testing); Test type: Non-Inferiority — The objective was to rule out a two-fold increase (non-inferiority testing) in the incidence rate of each of the maternal and infant adverse events, among vaccinated women with Boostrix and their infants as compared to the incidence in a matched cohort of unvaccinated women and their infants. The null hypothesis Ho: RR ≥ 2 was rejected if upper limit of the 98.75% CI for the adjusted RR was below 2; Risk Ratio (RR) = 1.38, 98.75% CI 2-sided [1.21 to 1.58] — Adjusted relative risk with 98.75% CI was estimated by Poisson regression model
Statistical Analysis 2: Comparison: Exposed Cohort women-on or After 1st Day of 27th Week of Pregnancy vs Unexposed Historical Cohort Women; Demonstration of adjusted RR for intra-uterine infections (chorioamnionitis and endometritis) in Exposed women cohort (on or after 1st day of 27th week of pregnancy) compared to Unexposed historical women cohort was less than 2 (non-inferiority testing); Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Risk Ratio (RR) = 1.28, 98.75% CI 2-sided [1.12 to 1.47] — Adjusted relative risk with 98.75% CI was estimated by Poisson regression model

2. Primary Outcome: Incidence Rate (Per 1000 Persons) of Prespecified Maternal Adverse Events for Exposed Cohort women-on or After 1st Day of 27th Week of Pregnancy and Unexposed Historical Cohort Women Groups
Description: Incidence rate (per 1000) consisted of the total number of adverse events in the numerator and the number of persons at risk in the denominator. Every unexposed woman was assigned an index date that is determined by the number of days from pregnancy start to the Boostrix vaccination date of her matched exposed woman. The same number of days calculated in the exposed woman was added to the pregnancy start of the unexposed woman to identify her index date. The pre-specified maternal adverse event assessed was preterm delivery.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Events per 1000 persons
Arm/Group | Exposed Cohort women-on or After 1st Day of 27th Week of Pregnancy | Unexposed Historical Cohort Women
Number analyzed (Participants) | 15767 | 15551
Events per 1000 persons | 64.63 [60.90 to 68.58] | 92.28 [87.84 to 96.94]
Statistical Analysis 1: Comparison: Exposed Cohort women-on or After 1st Day of 27th Week of Pregnancy vs Unexposed Historical Cohort Women; Demonstration of adjusted RR for preterm delivery in Exposed women cohort (on or after 1st day of 27th week of pregnancy) compared to Unexposed historical women cohort was less than 2 (non-inferiority testing); Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Risk Ratio (RR) = 0.71, 98.75% CI 2-sided [0.64 to 0.78] — Adjusted relative risk with 98.75% CI was estimated by Poisson regression model

3. Primary Outcome: Incidence Rate (Per 1000 Persons) of Pre-specified Infant Adverse Events for Exposed Cohort infants-on or After 1st Day of 27th Week of Pregnancy and Unexposed Historical Cohort Infants Groups
Description: The incidence rate (per 1000) of adverse events was calculated as the total number of adverse events in the numerator and the total of persons at risk in the denominator. The pre-specified infant adverse event assessed was small for gestational age.
Time Frame: From birth through 6 months of age
Population: The analysis was performed on live singleton infants for whom the event could be assessed and who born to women from Exposed cohort women-on or after 1st day of 27th week of pregnancy group and Unexposed historical cohort women group, who met eligibility criteria.
Measure: Number (95% Confidence Interval); unit: Events per 1000 persons
Arm/Group | Exposed Cohort infants-on or After 1st Day of 27th Week of Pregnancy | Unexposed Historical Cohort Infants
Number analyzed (Participants) | 15892 | 15626
Events per 1000 persons | 80.42 [76.30 to 84.76] | 75.00 [70.98 to 79.25]
Statistical Analysis 1: Comparison: Exposed Cohort infants-on or After 1st Day of 27th Week of Pregnancy vs Unexposed Historical Cohort Infants; Demonstration of adjusted RR for small for gestational age in Exposed infants cohort (on or after 1st day of 27th week of pregnancy) compared to Unexposed historical infants cohort was less than 2 (non-inferiority testing); Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Risk Ratio (RR) = 1.04, 98.75% CI 2-sided [0.94 to 1.16] — Adjusted RR with 98.75% CI-Poisson regression model

4. Secondary Outcome: Incidence Rate (Per 1000 Person-years) of Other Maternal Adverse Events for Exposed Cohort women-on or After 1st Day of 27th Week of Pregnancy and Unexposed Historical Cohort Women Groups
Description: The incidence rate (per 1000) of other maternal adverse events was calculated as the total number of adverse events in the numerator and the total person-years at risk in the denominator. Every unexposed woman was assigned an index date that is determined by the number of days from pregnancy start to the Boostrix vaccination date of her matched exposed woman. The same number of days calculated in the exposed woman was added to the pregnancy start of the unexposed woman to identify her index date. The analysis was used for hypothesis generation/signal detection, hence without adjustment for multiple comparisons. The other maternal adverse events assessed were poor fetal growth; placental abruption; preterm pre-labor rupture of membranes; maternal death.
Time Frame: as for outcome 1
Population: The analysis was performed on all women from the Exposed cohort women-on or after 1st day of 27th week of pregnancy group and the Unexposed historical cohort women group, who met the eligibility criteria and for whom the event could be assessed. Incidence rate of maternal death was not calculated for Unexposed Historical Cohort Women Group as none were reported in this group.
Measure: Number (95% Confidence Interval); unit: Events per 1000 persons-year
Arm/Group | Exposed Cohort women-on or After 1st Day of 27th Week of Pregnancy | Unexposed Historical Cohort Women
Number analyzed (Participants) | 16606 | 16606
Events per 1000 persons-year
  Poor fetal growth | 116.00 [103.99 to 129.40] | 137.63 [124.29 to 152.40]
  Placental abruption | 56.63 [48.45 to 66.19] | 44.59 [37.30 to 53.32]
  Preterm pre-labor rupture of membranes: number analyzed (Participants) | 16022 | 16022
  Preterm pre-labor rupture of membranes | 115.53 [103.52 to 128.94] | 141.52 [127.95 to 156.53]
  Maternal death: number analyzed (Participants) | 16606 | 0
  Maternal death | 0.43 [0.11 to 1.72] |
Statistical Analysis 1: Comparison: Exposed Cohort women-on or After 1st Day of 27th Week of Pregnancy vs Unexposed Historical Cohort Women; Assessment of adjusted RR for poor fetal growth in the Exposed pregnant women cohort (on or after 1st day of 27th week of pregnancy) compared to the Unexposed historical women cohort was 1 or differed from 1 (superiority testing); Test type: Superiority — The objective was to explore differences (superiority testing) in the incidence rate of each of the maternal and infant adverse events, among vaccinated women with Boostrix and their infants as compared to the incidence in a matched cohort of unvaccinated women and their infants. Superiority to be concluded if lower limit of the 95% CI for the adjusted RR is above 1; Risk Ratio (RR) = 0.83, 95% CI 2-sided [0.70 to 0.98] — Adjusted RR with 95% CI -Poisson regression model
Statistical Analysis 2: Comparison: Exposed Cohort women-on or After 1st Day of 27th Week of Pregnancy vs Unexposed Historical Cohort Women; Assessment of adjusted RR for placental abortion in Exposed women cohort (on or after 1st day of 27th week of pregnancy) compared to Unexposed historical women cohort was 1 or differed from 1 (superiority testing); Test type: Superiority — [test comment as in outcome 4, analysis 1]; Risk Ratio (RR) = 1.31, 95% CI 2-sided [0.99 to 1.72] — Adjusted RR with 95% CI - Poisson regression model
Statistical Analysis 3: Comparison: Exposed Cohort women-on or After 1st Day of 27th Week of Pregnancy vs Unexposed Historical Cohort Women; Assessment of adjusted RR for preterm pre-labor rupture of membranes in Exposed women cohort (on or after 1st day of 27th week of pregnancy) compared to Unexposed historical women cohort was 1 or differed from 1 (superiority testing); Test type: Superiority — [test comment as in outcome 4, analysis 1]; Risk Ratio (RR) = 0.76, 95% CI 2-sided [0.64 to 0.91] — Adjusted RR with 95% CI-Poisson regression model

5. Secondary Outcome: Incidence Rate (Per 1000 Persons) of Other Maternal Adverse Events for Exposed Cohort women-on or After 1st Day of 27th Week of Pregnancy and Unexposed Historical Cohort Women Groups
Description: The incidence rate (per 1000) consisted of the total number of adverse events in the numerator and the number of persons at risk in the denominator. Every unexposed woman was assigned an index date that is determined by the number of days from pregnancy start to the Boostrix vaccination date of her matched exposed woman. The same number of days calculated in the exposed woman was added to the pregnancy start of the unexposed woman to identify her index date. The analysis was used for hypothesis generation/signal detection, hence without adjustment for multiple comparisons. The other maternal adverse events assessed were stillbirth/fetal death; stillbirth/fetal death with congenital anomalies; transfusion during delivery hospitalization.
Time Frame: as for outcome 1
Population: The analysis was performed on all women from the Exposed cohort women-on or after 1st day of 27th week of pregnancy group and the Unexposed historical cohort women group, who met the eligibility criteria and for whom the specified event could be assessed. Incidence rate of stillbirth/fetal death with congenital anomalies was not calculated for Exposed Cohort women-on or After 1st Day of 27th Week of Pregnancy and Unexposed Historical Cohort Women Groups as none were reported in these groups.
Measure: Number (95% Confidence Interval); unit: Events per 1000 persons
Arm/Group | Exposed Cohort women-on or After 1st Day of 27th Week of Pregnancy | Unexposed Historical Cohort Women
Number analyzed (Participants) | 16368 | 16166
Events per 1000 persons
  Stillbirth/fetal death | 1.41 [0.93 to 2.11] | 2.41 [1.76 to 3.30]
  Stillbirth/fetal death with congenital anomalies: number analyzed (Participants) | 0 | 0
  Transfusion during delivery hospitalization: number analyzed (Participants) | 16335 | 16062
  Transfusion during delivery hospitalization | 12.79 [11.17 to 14.65] | 12.02 [10.43 to 13.84]
Statistical Analysis 1: Comparison: Exposed Cohort women-on or After 1st Day of 27th Week of Pregnancy vs Unexposed Historical Cohort Women; Assessment of adjusted RR for stillbirth/fetal death in Exposed women cohort (on or after 1st day of 27th week of pregnancy) compared to Unexposed historical women cohort was 1 or differed from 1 (superiority testing); Test type: Superiority — The objective was to explore differences (superiority testing) in the incidence rate of each of the maternal and infant adverse events, among vaccinated women with Boostrix and their infants as compared to the incidence in a matched cohort of unvaccinated women and their infants. The null hypothesis H0 RR =1 was rejected if lower limit of 95% CI for adjusted RR was above 1; Risk Ratio (RR) = 0.38, 95% CI 2-sided [0.22 to 0.67] — Adjusted RR with 95% CI-Poisson regression model
Statistical Analysis 2: Comparison: Exposed Cohort women-on or After 1st Day of 27th Week of Pregnancy vs Unexposed Historical Cohort Women; Assessment of adjusted RR for transfusion during delivery hospitalization in Exposed women cohort (on or after 1st day of 27th week of pregnancy) compared to Unexposed historical women cohort was 1 or differed from 1 (superiority testing); Test type: Superiority — The objective was to explore differences (superiority testing) in the incidence rate of each of the maternal and infant adverse events, among vaccinated women with Boostrix and their infants as compared to the incidence in a matched cohort of unvaccinated women and their infants. The null hypothesis H0 RR=1 was rejected if lower limit of 95% CI for adjusted RR was above 1; Risk Ratio (RR) = 1.07, 95% CI 2-sided [0.86 to 1.33] — Adjusted RR with 95% CI-Poisson regression model

6. Secondary Outcome: Incidence Rate (Per 1000 Persons) of Other Infant Adverse Events for Exposed Cohort infants-on or After 1st Day of 27th Week of Pregnancy and Unexposed Historical Cohort Infants Groups
Description: The incidence rate (per 1000) of other infant adverse events was calculated as the total number of adverse events in the numerator and the total of persons at risk in the denominator. The analysis was used for hypothesis generation/signal detection, hence without adjustment for multiple comparisons. The other infant adverse events assessed were neonatal death, congenital anomalies of: nervous system; eye; ear, face, or neck; cardiovascular system; respiratory system; clefts; upper gastrointestinal system; lower gastrointestinal system; genital organs; renal system; musculoskeletal system; limb; integument; other and unspecified.
Time Frame: From birth through 6 months of age
Population: The analysis was performed on live singleton infants for whom the specified event could be assessed, and who born to women from Exposed cohort women-on or after 1st day of 27th week of pregnancy group and Unexposed historical cohort women group, who met the eligibility criteria.
Measure: Number (95% Confidence Interval); unit: Events per 1000 persons
Arm/Group | Exposed Cohort infants-on or After 1st Day of 27th Week of Pregnancy | Unexposed Historical Cohort Infants
Number analyzed (Participants) | 16350 | 16088
Events per 1000 persons
  Neonatal death | 0.92 [0.55 to 1.52] | 1.06 [0.66 to 1.70]
  Congenital anomalies of nervous system | 2.81 [2.11 to 3.76] | 2.36 [1.72 to 3.25]
  Congenital anomalies of eye | 69.85 [66.05 to 73.87] | 60.48 [56.91 to 64.28]
  Congenital anomalies of ear, face, or neck | 16.27 [14.43 to 18.35] | 8.14 [6.86 to 9.66]
  Congenital anomalies of cardiovascular system | 24.40 [22.15 to 26.89] | 21.82 [19.67 to 24.20]
  Congenital anomalies of respiratory system | 13.76 [12.08 to 15.68] | 10.32 [8.86 to 12.01]
  Clefts | 1.96 [1.38 to 2.77] | 1.49 [1.00 to 2.23]
  Congenital anomalies of upper gastrointestinal system | 67.83 [64.08 to 71.79] | 37.85 [35.02 to 40.92]
  Congenital anomalies of lower gastrointestinal system | 1.35 [0.89 to 2.04] | 2.30 [1.67 to 3.17]
  Congenital anomalies of genital organs | 21.71 [19.57 to 24.09] | 18.46 [16.48 to 20.68]
  Congenital anomalies of renal system | 7.83 [6.58 to 9.31] | 5.91 [4.83 to 7.22]
  Congenital anomalies of musculoskeletal system | 16.27 [14.43 to 18.35] | 10.63 [9.15 to 12.35]
  Congenital anomalies of limb | 7.09 [5.91 to 8.51] | 6.90 [5.73 to 8.31]
  Congenital anomalies of integument | 58.04 [54.57 to 61.74] | 29.65 [27.14 to 32.39]
  Other and unspecified congenital anomalies | 1.96 [1.38 to 2.77] | 2.05 [1.46 to 2.89]
Statistical Analysis 1: Comparison: Exposed Cohort infants-on or After 1st Day of 27th Week of Pregnancy vs Unexposed Historical Cohort Infants; Assessment of adjusted RR for neonatal death in Exposed infants cohort (on or after 1st day of 27th week of pregnancy) compared to Unexposed historical infants cohort was 1 or differed from 1 (superiority testing); Test type: Superiority — [test comment as in outcome 5, analysis 2]; Risk Ratio (RR) = 0.81, 95% CI 2-sided [0.38 to 1.73] — Adjusted RR with 95% CI-Poisson regression model
Statistical Analysis 2: Comparison: Exposed Cohort infants-on or After 1st Day of 27th Week of Pregnancy vs Unexposed Historical Cohort Infants; Assessment of adjusted RR for congenital anomalies of nervous system in Exposed infants cohort (on or after 1st day of 27th week of pregnancy) compared to Unexposed historical infants cohort was 1 or differed from 1 (superiority testing); Test type: Superiority — [test comment as in outcome 5, analysis 2]; Risk Ratio (RR) = 1.35, 95% CI 2-sided [0.81 to 2.24] — Adjusted RR with 95% CI-Poisson regression model
Statistical Analysis 3: Comparison: Exposed Cohort infants-on or After 1st Day of 27th Week of Pregnancy vs Unexposed Historical Cohort Infants; Assessment of adjusted RR for congenital anomalies of eye in Exposed infants cohort (on or after 1st day of 27th week of pregnancy) compared to Unexposed historical infants cohort was 1 or differed from 1 (superiority testing); Test type: Superiority — [test comment as in outcome 5, analysis 2]; Risk Ratio (RR) = 1.17, 95% CI 2-sided [1.06 to 1.29] — Adjusted RR with 95% CI-Poisson regression model
Statistical Analysis 4: Comparison: Exposed Cohort infants-on or After 1st Day of 27th Week of Pregnancy vs Unexposed Historical Cohort Infants; Assessment of adjusted RR for congenital anomalies of ear, face or neck in Exposed infants cohort (on or after 1st day of 27th week of pregnancy) compared to Unexposed historical infants cohort was 1 or differed from 1 (superiority testing; Test type: Superiority — [test comment as in outcome 5, analysis 2]; Risk Ratio (RR) = 2.02, 95% CI 2-sided [1.59 to 2.55] — Adjusted RR with 95% CI-Poisson regression model
Statistical Analysis 5: Comparison: Exposed Cohort infants-on or After 1st Day of 27th Week of Pregnancy vs Unexposed Historical Cohort Infants; Assessment of adjusted RR for congenital anomalies of cardiovascular system in Exposed infants cohort (on or after 1st day of 27th week of pregnancy) compared to Unexposed historical infant cohort was 1 or differed from 1 (superiority testing); Test type: Superiority — [test comment as in outcome 5, analysis 2]; Risk Ratio (RR) = 1.12, 95% CI 2-sided [0.96 to 1.31] — Adjusted RR with 95% CI-Poisson regression model
Statistical Analysis 6: Comparison: Exposed Cohort infants-on or After 1st Day of 27th Week of Pregnancy vs Unexposed Historical Cohort Infants; Assessment of adjusted RR for congenital anomalies of respiratory system in Exposed infants cohort (on or after 1st day of 27th week of pregnancy) compared to Unexposed historical infants cohort was1 or differed from 1 (superiority testing); Test type: Superiority — [test comment as in outcome 5, analysis 2]; Risk Ratio (RR) = 1.34, 95% CI 2-sided [1.07 to 1.68] — Adjusted RR with 95% CI-Poisson regression model
Statistical Analysis 7: Comparison: Exposed Cohort infants-on or After 1st Day of 27th Week of Pregnancy vs Unexposed Historical Cohort Infants; Assessment of adjusted RR for clefts in Exposed infants cohort (on or after 1st day of 27th week of pregnancy) compared to Unexposed historical infants cohort was 1 or differed from 1 (superiority testing); Test type: Superiority — [test comment as in outcome 5, analysis 2]; Risk Ratio (RR) = 1.41, 95% CI [0.78 to 2.57] — Adjusted RR with 95% CI-Poisson regression model
Statistical Analysis 8: Comparison: Exposed Cohort infants-on or After 1st Day of 27th Week of Pregnancy vs Unexposed Historical Cohort Infants; Assessment of adjusted RR for congenital anomalies of upper gastrointestinal system in Exposed infants cohort (on or after 1st day of 27th week of pregnancy) compared to Unexposed historical infants cohort was 1 or differed from 1 (superiority testing); Test type: Superiority — [test comment as in outcome 5, analysis 2]; Risk Ratio (RR) = 1.75, 95% CI 2-sided [1.57 to 1.95] — Adjusted RR with 95% CI-Poisson regression model
Statistical Analysis 9: Comparison: Exposed Cohort infants-on or After 1st Day of 27th Week of Pregnancy vs Unexposed Historical Cohort Infants; Assessment of adjusted RR for congenital anomalies of lower gastrointestinal system in Exposed infants cohort (on or after 1st day of 27th week of pregnancy) compared to Unexposed historical infants cohort was 1 or differed from 1 (superiority testing); Test type: Superiority — [test comment as in outcome 5, analysis 2]; Risk Ratio (RR) = 0.63, 95% CI 2-sided [0.36 to 1.12] — Adjusted RR with 95% CI-Poisson regression model
Statistical Analysis 10: Comparison: Exposed Cohort infants-on or After 1st Day of 27th Week of Pregnancy vs Unexposed Historical Cohort Infants; Assessment of adjusted RR for congenital anomalies of genital organs in Exposed infants cohort (on or after 1st day of 27th week of pregnancy) compared to Unexposed historical infants cohort was 1 or differed from 1 (superiority testing); Test type: Superiority — [test comment as in outcome 5, analysis 2]; Risk Ratio (RR) = 1.19, 95% CI 2-sided [1.01 to 1.42] — Adjusted RR with 95% CI-Poisson regression model
Statistical Analysis 11: Comparison: Exposed Cohort infants-on or After 1st Day of 27th Week of Pregnancy vs Unexposed Historical Cohort Infants; Assessment of adjusted RR for congenital anomalies of renal system in Exposed infants cohort (on or after 1st day of 27th week of pregnancy) compared to Unexposed historical infants cohort was 1 or differed from 1 (superiority testing; Test type: Superiority — [test comment as in outcome 5, analysis 2]; Risk Ratio (RR) = 1.40, 95% CI 2-sided [1.04 to 1.88] — Adjusted RR with 95% CI-Poisson regression model
Statistical Analysis 12: Comparison: Exposed Cohort infants-on or After 1st Day of 27th Week of Pregnancy vs Unexposed Historical Cohort Infants; Assessment of adjusted RR for congenital anomalies of musculoskeletal system in Exposed infants cohort (on or after 1st day of 27th week of pregnancy) compared to Unexposed historical infants cohort was 1 or differed from 1 (superiority testing); Test type: Superiority — [test comment as in outcome 5, analysis 2]; Risk Ratio (RR) = 1.50, 95% CI [1.21 to 1.86] — Adjusted RR with 95% CI-Poisson regression model
Statistical Analysis 13: Comparison: Exposed Cohort infants-on or After 1st Day of 27th Week of Pregnancy vs Unexposed Historical Cohort Infants; Assessment of adjusted RR for congenital anomalies of limb in Exposed infants cohort (on or after 1st day of 27th week of pregnancy) compared to Unexposed historical infants cohort was 1 or differed from 1 (superiority testing); Test type: Superiority — [test comment as in outcome 5, analysis 2]; Risk Ratio (RR) = 1.13, 95% CI 2-sided [0.85 to 1.52] — Adjusted RR with 95% CI-Poisson regression model
Statistical Analysis 14: Comparison: Exposed Cohort infants-on or After 1st Day of 27th Week of Pregnancy vs Unexposed Historical Cohort Infants; Assessment of adjusted RR for congenital anomalies of integument in Exposed infants cohort (on or after 1st day of 27th week of pregnancy) compared to Unexposed historical infants cohort was 1 or differed from 1 (superiority testing); Test type: Superiority — [test comment as in outcome 5, analysis 2]; Risk Ratio (RR) = 1.98, 95% CI 2-sided [1.76 to 2.23] — Adjusted RR with 95% CI-Poisson regression model
Statistical Analysis 15: Comparison: Exposed Cohort infants-on or After 1st Day of 27th Week of Pregnancy vs Unexposed Historical Cohort Infants; Assessment of adjusted RR for other and unspecified congenital anomalies in Exposed infants cohort (on or after 1st day of 27th week of pregnancy) compared to Unexposed historical infants cohort was 1 or differed from 1 (superiority testing); Test type: Superiority — [test comment as in outcome 5, analysis 2]; Risk Ratio (RR) = 1.09, 95% CI 2-sided [0.64 to 1.85] — Adjusted RR with 95% CI-Poisson regression model

7. Secondary Outcome: Incidence Rate (Per 1000 Person-years) of Women Adverse Events for Exposed Cohort Women-before 1st Day of 27th Week of Pregnancy Group
Description: The incidence rate (per 1000) was calculated as the total number of adverse events in the numerator and the total person-years at risk in the denominator. Due to the small sample size, the analysis of these women adverse events was descriptive. The women adverse events assessed were pre-eclampsia and eclampsia; intra-uterine infections; poor fetal growth; placental abruption; preterm pre-labor rupture of membranes; maternal death.
Time Frame: For the Exposed cohort women-before 1st day of 27th week of pregnancy: from date of Boostrix vaccination until end of enrollment or pregnancy, whichever came first, up to 40 weeks
Population: The analysis was performed on women from Exposed cohort women-before 1st day of 27th week of pregnancy group who met the eligibility criteria and for whom the specified event could be assessed. Incidence rate of placental abruption and maternal death was not calculated for Exposed Cohort Women-before 1st Day of 27th Week of Pregnancy Group as none were reported in this group.
Measure: Number (95% Confidence Interval); unit: Events per 1000 persons-year
Arm/Group | Exposed Cohort Women-before 1st Day of 27th Week of Pregnancy
Number analyzed (Participants) | 65
Events per 1000 persons-year
  Pre-eclampsia and eclampsia | 354.50 [146.26 to 755.09]
  Intra-uterine infections | 176.42 [45.85 to 525.92]
  Poor fetal growth | 119.75 [20.81 to 453.17]
  Placental abruption: number analyzed (Participants) | 0
  Preterm pre-labor rupture of membranes | 117.65 [20.45 to 445.22]
  Maternal death: number analyzed (Participants) | 0

8. Secondary Outcome: Incidence Rate (Per 1000 Persons) of Women Adverse Events Presented for Exposed Cohort Women-before 1st Day of 27th Week of Pregnancy Group
Description: The incidence rate (per 1000) consisted of the total number of adverse events in the numerator and the number of persons at risk in the denominator. The adverse events of this analysis include the adverse events presented in the above outcomes as well as spontaneous and therapeutic abortion with or without congenital anomalies in pregnant women vaccinated with Boostrix before the 27th week of gestation. Due to the small sample size, the analysis of these women adverse events was descriptive. The women adverse events assessed were stillbirth/fetal death; stillbirth/fetal death with congenital anomalies; spontaneous abortion; spontaneous abortion with congenital anomalies; therapeutic abortion; therapeutic abortion with congenital anomalies; transfusion during delivery hospitalization; preterm delivery.
Time Frame: as for outcome 7
Population: The analysis was performed on women from Exposed cohort women-before 1st day of 27th week of pregnancy group who met the eligibility criteria and for whom the specified event could be assessed. Incidence rate of stillbirth/fetal death, stillbirth/fetal death with congenital anomalies, spontaneous abortion with congenital anomalies, therapeutic abortion, or therapeutic abortion with congenital anomalies was not calculated for the analyzed group as none were reported in this group.
Measure: Number (95% Confidence Interval); unit: Events per 1000 persons
Arm/Group | Exposed Cohort Women-before 1st Day of 27th Week of Pregnancy
Number analyzed (Participants) | 65
Events per 1000 persons
  Stillbirth/fetal death: number analyzed (Participants) | 0
  Stillbirth/fetal death with congenital anomalies: number analyzed (Participants) | 0
  Spontaneous abortion | 15.38 [0.80 to 94.03]
  Spontaneous abortion with congenital anomalies: number analyzed (Participants) | 0
  Therapeutic abortion: number analyzed (Participants) | 0
  Therapeutic abortion with congenital anomalies: number analyzed (Participants) | 0
  Transfusion during delivery hospitalization: number analyzed (Participants) | 64
  Transfusion during delivery hospitalization | 15.63 [0.82 to 95.41]
  Preterm delivery: number analyzed (Participants) | 64
  Preterm delivery | 46.88 [12.18 to 139.59]

9. Secondary Outcome: Incidence Rate (Per 1000 Persons) of Infant Adverse Events for Exposed Cohort Infants-before 1st Day of 27th Week of Pregnancy Group
Description: The incidence rate (per 1000) was calculated as the total number of adverse events in the numerator and the total of persons at risk in the denominator. The adverse events of this analysis include adverse events presented in the above outcomes, among the infants whose mothers were vaccinated with Boostrix before the 27th week of gestation. Due to the small sample size, the analysis of these infant adverse events was descriptive. The infant adverse events assessed were: small for gestational age; neonatal death; congenital anomalies of: nervous system; eye; ear, face, or neck; cardiovascular system; respiratory system; clefts; upper gastrointestinal system; lower gastrointestinal system; genital organs; renal system; musculoskeletal system; limb; integument; other and unspecified.
Time Frame: From birth through 6 months of age
Population: The analysis was performed on infants for whom the specified event could be assessed, who were born to women from Exposed cohort women-before 1st day of 27th week of pregnancy group, and who met the eligibility criteria. Incidence rate of neonatal death; clefts; congenital anomalies of: nervous system, respiratory system; lower gastrointestinal system, limb, or other and unspecified congenital anomalies was not calculated for the analyzed group as none were reported in this group.
Measure: Number (95% Confidence Interval); unit: Events per 1000 persons
Arm/Group | Exposed Cohort Infants-before 1st Day of 27th Week of Pregnancy
Number analyzed (Participants) | 68
Events per 1000 persons
  Small for gestational age: number analyzed (Participants) | 60
  Small for gestational age | 116.67 [52.10 to 231.77]
  Neonatal death: number analyzed (Participants) | 0
  Clefts: number analyzed (Participants) | 0
  Congenital anomalies of nervous system: number analyzed (Participants) | 0
  Congenital anomalies of eye | 88.24 [36.38 to 188.56]
  Congenital anomalies of ear, face, or neck | 73.53 [27.39 to 170.21]
  Congenital anomalies of cardiovascular system | 14.71 [0.77 to 90.12]
  Congenital anomalies of respiratory system: number analyzed (Participants) | 0
  Congenital anomalies of upper gastrointestinal system | 14.71 [0.77 to 90.12]
  Congenital anomalies of lower gastrointestinal system: number analyzed (Participants) | 0
  Congenital anomalies of genital organs | 44.12 [11.46 to 131.90]
  Congenital anomalies of renal system | 14.71 [0.77 to 90.12]
  Congenital anomalies of musculoskeletal system | 14.71 [0.77 to 90.12]
  Congenital anomalies of limb: number analyzed (Participants) | 0
  Congenital anomalies of integument | 102.94 [45.87 to 206.51]
  Other and unspecified congenital anomalies: number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: For each woman from date of Boostrix vaccination (Exposed cohort women-on or after 1st day of 27th week of pregnancy Group and Exposed cohort women-before 1st day of 27th week of pregnancy Group), and from an index date (Unexposed historical cohort women) until end of enrollment (up to 13 weeks) or pregnancy (up to 40 weeks). For infants, from birth through 6 months of age.
Description: Classification of events as SAE/other AE is unknown, all events were reported in SAE section. SAEs data was collected from different analytic populations for whom the event could be evaluated. Therefore for: Preterm delivery, Preterm pre-labor rupture of membranes, Stillbirths/fetal deaths without congenital anomalies, Transfusion during delivery hospitalization, Small for gestational age, the number of participants at risk differs from total number at risk for SAEs reported in all Arms.
Arm/Group | Exposed Cohort women-on or After 1st Day of 27th Week of Pregnancy | Unexposed Historical Cohort Women | Exposed Cohort Women-before 1st Day of 27th Week of Pregnancy | Exposed Cohort infants-on or After 1st Day of 27th Week of Pregnancy | Unexposed Historical Cohort Infants | Exposed Cohort Infants-before 1st Day of 27th Week of Pregnancy
All-Cause Mortality (participants affected / at risk) | 2/16606 | 0/16606 | 0/65 | 15/16350 | 17/16088 | 0/68
Serious Adverse Events (participants affected / at risk) | 3733/16606 | 3679/16606 | 18/65 | 5540/16350 | 4211/16088 | 30/68
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Exposed Cohort women-on or After 1st Day of 27th Week of Pregnancy (N=16606) | Unexposed Historical Cohort Women (N=16606) | Exposed Cohort Women-before 1st Day of 27th Week of Pregnancy (N=65) | Exposed Cohort infants-on or After 1st Day of 27th Week of Pregnancy (N=16350) | Unexposed Historical Cohort Infants (N=16088) | Exposed Cohort Infants-before 1st Day of 27th Week of Pregnancy (N=68)
Preeclampsia/eclampsia (General disorders) | 874 (874) | 588 (588) | 6 (6) | 0/0 (0) | 0/0 (0) | 0/0 (0) — No medical dictionary coding applied to this event
Intra-uterine infections (General disorders) | 811 (811) | 558 (558) | 3 (3) | 0/0 (0) | 0/0 (0) | 0/0 (0) — No medical dictionary coding applied to this event
Small for gestational age (General disorders) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 1278/15892 (1278) | 1172/15626 (1172) | 7/60 (7) — No medical dictionary coding applied to this event
Preterm delivery (General disorders) | 1019/15767 (1019) | 1435/15551 (1435) | 3/64 (3) | 0/0 (0) | 0/0 (0) | 0/0 (0) — No medical dictionary coding applied to this event
Transfusion during delivery hospitalization (General disorders) | 209/16335 (209) | 193/16062 (193) | 1/64 (1) | 0/0 (0) | 0/0 (0) | 0/0 (0) — No medical dictionary coding applied to this event
Poor fetal growth (General disorders) | 320 (320) | 368 (368) | 2 (2) | 0/0 (0) | 0/0 (0) | 0/0 (0) — No medical dictionary coding applied to this event
Placental abruption (General disorders) | 157 (157) | 120 (120) | 0 (0) | 0/0 (0) | 0/0 (0) | 0/0 (0) — No medical dictionary coding applied to this event
Preterm pre-labor rupture of membranes (General disorders) | 318/16022 (318) | 378/16022 (378) | 2 (2) | 0/0 (0) | 0/0 (0) | 0/0 (0) — No medical dictionary coding applied to this event
Congenital anomalies of nervous system (General disorders) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 46 (46) | 38 (38) | 0 (0) — No medical dictionary coding applied to this event
Congenital anomalies of eye (General disorders) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 1142 (1142) | 973 (973) | 6 (6) — No medical dictionary coding applied to this event
Congenital anomalies of ear, face or neck (General disorders) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 266 (266) | 131 (131) | 5 (5) — No medical dictionary coding applied to this event
Congenital anomalies of cardiovascular system (General disorders) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 399 (399) | 351 (351) | 1 (1) — No medical dictionary coding applied to this event
Congenital anomalies of respiratory system (General disorders) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 225 (225) | 166 (166) | 0 (0) — No medical dictionary coding applied to this event
Clefts (General disorders) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 32 (32) | 24 (24) | 0 (0) — No medical dictionary coding applied to this event
Congenital anomalies of upper gastrointestinal system (General disorders) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 1109 (1109) | 609 (609) | 1 (1) — No medical dictionary coding applied to this event
Congenital anomalies of lower gastrointestinal system (General disorders) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 22 (22) | 37 (37) | 0 (0) — No medical dictionary coding applied to this event
Congenital anomalies of genital organs (General disorders) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 355 (355) | 297 (297) | 3 (3) — No medical dictionary coding applied to this event
Congenital anomalies of renal system (General disorders) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 128 (128) | 95 (95) | 1 (1) — No medical dictionary coding applied to this event
Congenital anomalies of musculoskeletal system (General disorders) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 266 (266) | 171 (171) | 1 (1) — No medical dictionary coding applied to this event
Congenital anomalies of limb (General disorders) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 116 (116) | 111 (111) | 0 (0) — No medical dictionary coding applied to this event
Congenital anomalies of integument (General disorders) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 949 (949) | 477 (477) | 7 (7) — No medical dictionary coding applied to this event
Other and unspecified congenital anomalies (General disorders) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 32 (32) | 33 (33) | 0 (0) — No medical dictionary coding applied to this event
Spontaneous abortion (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0/0 (0) | 0/0 (0) | 0/0 (0) — No medical dictionary coding applied to this event
Maternal deaths (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0/0 (0) | 0/0 (0) | 0/0 (0) — No medical dictionary coding applied to this event
Stillbirths/fetal deaths without congenital anomalies (General disorders) | 23/16368 (23) | 39/16166 (39) | 0 (0) | 0/0 (0) | 0/0 (0) | 0/0 (0) — No medical dictionary coding applied to this event
Neonatal deaths (General disorders) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 15 (15) | 17 (17) | 0 (0) — No medical dictionary coding applied to this event

LIMITATIONS AND CAVEATS:
Main limitation: difference in background rates and time periods for both cohorts. Other: confounding by indication possible for a less select historical unvaccinated population. The study wasn't designed to study safety of exposure before 27 weeks of gestation and was conducted in a prepaid health plan, so findings may not be generalized to uninsured populations. Congenital anomalies analysis performed by event code without adjustment for multiple testing.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2019-11-12): https://cdn.clinicaltrials.gov/large-docs/77/NCT03463577/Prot_000.pdf
  • Statistical Analysis Plan (2019-12-02): https://cdn.clinicaltrials.gov/large-docs/77/NCT03463577/SAP_001.pdf